CLINICAL TRIAL: NCT07039526
Title: Single Dose Investigator Initiated Pilot Study to Investigate CYTALUX (Pafolacianine) for Intraoperative Detection of Malignant Tissue in Subjects Undergoing Surgical Resection for Cancer.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: John Waters (Other)
Collaborators: On Target Laboratories, LLC (Industry)
Responsible Party: Sponsor-Investigator, John Waters, MD, Assistant Professor, Cardiothoracic Surgery, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU20250049
Record Dates: First submitted 2025-06-17; First posted 2025-06-26 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Cancer; Gastrointestinal Cancers; Gynecologic Cancers
Keywords: Pafolacianine; CYTALUX; Folate receptor-alpha; Near-infrared fluorescence imaging; Intraoperative imaging; Fluorescence-guided surgery; esophageal cancer; gastrointestinal cancer
MeSH Terms: conditions — Esophageal Neoplasms; Gastrointestinal Neoplasms | interventions — Pafolacianine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CYTALUX™ (pafolacianine) injection group (Experimental): Single arm study, every patient receives the study intervention.
  Interventions: Drug: CYTALUX™ (pafolacianine) injection preoperatively

INTERVENTIONS:
Drug: CYTALUX™ (pafolacianine) injection preoperatively — CYTALUX™ (pafolacianine) injection: folate analog ligand conjugated with an indole cyanine green-like dye as a solution in vials containing 1.6 mL at 2 mg/mL. Each subject will be administered a single intravenous dose of not less than 1 hours before and not more than 24 hours before initiation of intraoperative NIR fluorescent imaging.

SUMMARY:
The goal of clinical trial is to test an FDA approved drug called Pafolacianine that attaches to cancer cells and lights up when seen through a special camera system in adults with a suspected primary diagnosis, or a high clinical suspicion of gastrointestinal, fore gut, pancreatic, hepatobiliary, esophageal malignancies and gyn malignancies planned for HIPEC/debulking, warranting surgery. The main question it aims to answer is:

• Can CYTALUX™ (pafolacianine) injection used with near-infrared (NIR) fluorescent imaging improve the detection of malignant tissue in subjects undergoing surgical resection for cancer? Participants taking part in this study will receive the study medication. Then, during the surgery the investigator team will turn on the camera to evaluate if the tumor is visible with the help of the study medication. Taking part in this study will last about 2 months.

DETAILED DESCRIPTION:
Background and Rationale:

Gastroesophageal and pancreatic cancers are aggressive malignancies with limited curative options. Complete surgical resection (R0) remains the cornerstone of curative intent. However, current intraoperative tools-visual inspection, palpation, and endoscopy-are limited in accurately delineating tumor margins and detecting occult lesions. High recurrence rates after surgery suggest a need for improved intraoperative detection techniques.

Folate receptor-alpha (FRα) is overexpressed in a variety of epithelial tumors, including gastric and pancreatic cancers. Recent studies have demonstrated that over one-third of gastric cancers and a subset of peritoneal metastases from gastrointestinal tumors overexpress FRα, making them amenable to targeted imaging. Pafolacianine is a folate analog conjugated to a near-infrared fluorescent dye designed to bind to FRα, enabling real-time intraoperative visualization of cancerous tissue using NIR imaging systems.

Investigational Product:

CYTALUX™ (pafolacianine) is an intravenously administered imaging agent developed by On Target Laboratories, Inc. It consists of OTL0038, a folate analog conjugated to an indole-cyanine green-like dye. The agent selectively binds FRα and emits fluorescence in the NIR spectrum (excitation: 760-785 nm; emission: 790-815 nm), providing high-contrast imaging during surgery.

Mechanism of Action:

Following IV administration, pafolacianine distributes systemically and is cleared rapidly from normal tissues. In FRα-expressing tumor cells, the agent is retained due to receptor-mediated endocytosis. Upon NIR illumination, malignant tissues fluoresce, allowing surgeons to visualize tumors, metastatic nodules, and lymph nodes intraoperatively. This mechanism supports improved tumor localization, identification of positive margins, and enhanced detection of otherwise occult lesions.

Preclinical and Clinical Data:

Preclinical studies in KB human carcinoma cell lines and murine xenograft models have shown high binding affinity to FRα (KD = 10.4 nM) and specific tumor fluorescence. Safety evaluations in rats and dogs demonstrated no phototoxicity or systemic toxicity. Pafolacianine has been evaluated in completed Phase 1, 2, and 3 trials in ovarian and lung cancers (e.g., NCT03180307), where it identified additional malignant lesions or positive margins in 25-40% of patients, reinforcing its clinical utility.

Clinical Need and Future Application:

There is a substantial unmet need for real-time intraoperative tools that enhance surgical decision-making in gastrointestinal oncology. Pafolacianine offers potential benefits in:

Identifying primary and metastatic lesions in gastroesophageal and pancreatic cancer

Assessing peritoneal carcinomatosis in advanced gastric and appendiceal malignancies

Improving accuracy in cytoreductive surgeries and guiding HIPEC decisions

Given the expression profile of FRα in gastrointestinal and other epithelial malignancies, CYTALUX is anticipated to be beneficial for a broader spectrum of tumors beyond ovarian and lung cancers.

Imaging Protocol:

Participants will receive a single IV dose of pafolacianine prior to surgery. NIR imaging will be conducted intraoperatively using a compatible device. Fluorescent lesions will be documented and evaluated for correlation with histopathology. Standard-of-care surgical procedures (e.g., resection, lymphadenectomy) will proceed per usual protocol, supplemented by fluorescent signal guidance.

Endpoints:

Primary: Proportion of additional malignant lesions detected with NIR imaging not identified through standard visualization techniques.

Secondary: Rate of complete (R0) resections, correlation of fluorescence with histologically confirmed malignancy, adverse events related to pafolacianine administration.

Safety Considerations:

CYTALUX has demonstrated a favorable safety profile with no significant toxicity observed in preclinical or clinical settings. The agent is not associated with phototoxicity, and systemic clearance is rapid in non-target tissues.

ELIGIBILITY:
Inclusion Criteria:

1. Male and Female patients 18 years of age and older
2. Have a primary diagnosis, or a high clinical suspicion, of gastrointestinal, fore gut, pancreatic, hepatobiliary, esophageal malignancies and gyn malignancies planned for HIPEC/debulking, warranting surgery.
3. Are scheduled to undergo surgical intervention for tumor resection or diagnostic laparoscopy for assessment of disease burden.
4. Willingness to stop the use of folate, folic acid, or folate-containing supplements within 48 hours before administration of Cytalux
5. Willingness of research participant or legal guardian/representative to give written informed consent.

Exclusion Criteria:

1. Any medical condition that in the opinion of the investigators could potentially jeopardize the safety of the subject
2. History of anaphylactic reactions to products containing indocyanine green for near infrared imaging. Subjects with a medical history of 'idiopathic anaphylaxis' will require evaluation.
3. History of allergy to any of the components of CYTALUX™ (pafolacianine) injection
4. Presence of any psychological, familial, sociological condition or geographical challenges potentially hampering compliance with the study protocol or follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with one or more NIR fluorescence positive lesion not detected under normal light and/or palpation | Day 1 intra-operatively post intervention
  Proportion of subjects who have one or more NIR fluorescence positive lesion not detected under normal light and/or palpation will be measured in this outcome.

SECONDARY OUTCOMES:
Number of lesions that are simultaneously fluorescence positive and cancer positive | Day 1 intra-operatively post intervention
  NIR Imaging will take place at least 1 hour but no more than 24 hours after the end of the administration

CONTACTS AND LOCATIONS:
Overall Officials: John Waters, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Clemments University Hospital, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: OTL38 for Intra-operative Imaging of Folate Receptor Positive Ovarian Cancer — https://clinicaltrials.gov/study/NCT03180307?term=NCT03180307&rank=1